CLINICAL TRIAL: NCT03620630
Title: Evidence Generation for the Clinical Efficacy and Cost Effectiveness of myCOPD in Patients With Mild and Moderate Newly Diagnosed COPD
Brief Title: Clinical Efficacy and Cost Effectiveness of MYCOPD in Patients With Mild and Moderate Newly Diagnosed COPD
Acronym: EARLY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: my mhealth Ltd (Industry)
Collaborators: Innovate UK (Other Government); Imperial College London (Other); Hull University Teaching Hospitals NHS Trust (Other Government); Hampshire Hospitals NHS Foundation Trust (Other); Central London Community Healthcare NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MMH/RD/002
Record Dates: First submitted 2018-07-17; First posted 2018-08-08 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Randomised controlled Feasibility study
Who Masked: Outcomes Assessor
Masking Description: End of study visit to be completed by a blinded team
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients allocated to usual care will continue with their current NHS management in line with national and local guidelines.
- myCOPD (Active Comparator): Patients allocated to the myCOPD arm will receive access to a web based application called myCOPD
  Interventions: Device: myCOPD

INTERVENTIONS:
Device: myCOPD — myCOPD is a multi faceted web based application designed to support people with COPD in the Long term management of their COPD.
  Arms: myCOPD

SUMMARY:
Millions of patients in the UK live with long term medical conditions such as diabetes, heart disease and lung diseases. These conditions are the major cause of ill health in the UK and cost the NHS billions of pounds each year. One long term condition that carries an enormous impact for patients and the NHS is COPD (Chronic Obstructive Pulmonary Disease). This lung condition affects over one million patients in the UK and is one of the major causes of admission to hospital.

Involvement of patients in the management of their own medical conditions (self-care) has been shown to improve how individuals feel, reduce the frequency of medical emergencies and reduce the costs of health care. In order to self-care successfully patients require the correct knowledge, skills and the confidence to make the right decisions; about their treatments, use of healthcare services and lifestyle choices. Recently the use of digital tools such as apps and websites has been shown to help patients with self-care and thus to improve their health. However in the UK there are very few providers of apps that are fully accredited by the NHS and only one that has been fully funded to provide apps nationally.

My mhealth (short for my mobile health) is a UK company founded by NHS doctors which provides high quality digital tools (apps) to enable patients to access information about their condition and treatments and to record symptoms on their phones, tablets, computers or even smart TVs. MyMHealth has produced an app called MyCOPD which has been issued by the NHS to many thousands of patients in the UK. This was because it has been shown to improve the way patients with more severe COPD use their treatment and improved their day to day function through use of an online exercise programme.

In this proposed study the MyMHealth team will work with NHS professionals to explore how an app called MyCOPD could help patients with mild disease and particularly those newly diagnosed with the condition. Investigators will explore how these patients can use the app and whether it's use can improve the ability to self-manage their condition. Investigators will study the potential for the app to establish appropriate and active decision making by patients and the impact of this on the use of NHS resources and the costs of day to day care.

DETAILED DESCRIPTION:
COPD is a disabling, smoking related lung disease that is associated with symptoms of shortness of breath, cough and wheeze. The natural history is one of progressive decline, frequently punctuated by periods of rapid worsening termed acute exacerbations. The functional limitation experienced by individuals with COPD, their propensity to exacerbations and the high levels of psychological and physical co-morbidities place a significant burden on health and social care systems. It is estimated that COPD will become the 4th leading cause of death worldwide by 2030.

A typical UK city has over 7,500 patients with COPD on primary care registries and it is estimated that there are an additional 6,500 individuals living with the disease that have not yet been diagnosed. The NHS in England encourages opportunistic and systematic case finding to achieve early disease recognition. However, the merits of this approach are unclear due to a lack of evidence that early disease identification alters outcomes.

A recent randomised controlled trial undertaken in China has suggested that initiation of Tiotropium in patients with early disease may reduce the rate of lung function decline compared to placebo. This phenomenon was also observed in a subgroup analysis of young and milder COPD patients in the UPLIFT trial. Prior to these observations, smoking cessation was the only means of altering disease course in patients with early disease and there is conflicting evidence as to whether identifying COPD in smokers helps to achieve this or not. The possibility that early drug initiation may alter disease trajectory and improve long term health outcomes, makes early diagnosis appealing.

It is recognised that at the time of COPD diagnosis, patients are already less physically active than their peers that do not have airflow obstruction. This suggests that patients alter their behaviour to avoid symptoms before they perceive a problem significant enough to warrant medical attention. Physical inactivity is common in COPD patients and breathlessness is cited as the most common cause. Physical inactivity is one of the strongest predictors of death in COPD patients.To date, interventions that aim to increase physical activity have had limited success. This may be because interventions are targeted at patients with established disease when behaviour change is already established. We hypothesise that a better approach would be to prevent behaviour change in the first place rather than try to reverse it after it has occurred. Given the major barrier to physical activity is breathlessness and that this appears to impact individuals early in the disease, often before presentation, we propose that early intervention with therapies proven to reduce breathlessness will offer the greatest benefit.

Recent years have seen the development of new therapeutic strategies in COPD. A new class of inhaled therapy has emerged in the form of combined long acting beta-2 agonists (LABA) and long acting muscarinic receptor antagonists (LAMA). This dual bronchodilator approach achieves greater improvements in lung function, symptoms, quality of life and exacerbation frequency compared to the individual components alone. Early initiation of therapy with dual bronchodilation has the potential to prevent the reduction in physical activity that occurs due to exertional breathlessness and is now advocated as the first line treatment for COPD.

Therefore there is an increased need to explore strategies to support patients with mild, moderate and early COPD as the rationale for treatment develops. Here the evidence that self-management can play an important contribution to improving clinical outcomes whilst reducing health care resource use and associated costs is great. In order to effectively self-manage, patients require the knowledge, skills and confidence to make appropriate decisions about their care. When newly diagnosed, there are very few opportunities for patients to learn about their condition and develop the skills to case manage effectively. Consequently patients with LTC's often rely on health care professional to guide them and are unaware of appropriator measures they can take themselves to improve their own health. The use of digital technologies, particularly apps has been suggested as a way of empowering patients to self-manage effectively. The provision of high quality information and advice on medication, health promoting activities and improvements in adherence via apps can help patient gain the skills and confidence they need to effectively manage their conditions.

MyMHealth is a leading digital health provider that is one of the very few MHRA approved app developers and the only provider to be funded by NHS England through the National Innovation and Technology Tariff to provide patients with high quality apps to help them manage their health. MyCOPD is such a patient platform and the NHS and NICE approvals have led to the distribution of access licenses to over 50 000 patients with COPD in England. This product is therefore at the vanguard of the digital health revolution in the UK based on a strong evidence base of benefit in patient with established and more severe disease. However the majority of patients with COPD have milder disease and currently patients with mild to moderate or newly diagnosed COPD are not funded to receive the app as part of their routine care as the evidence base for its use is not mature. This study seeks to explore the potential for the use of MyCOPD to improve COPD patients' activation, disease knowledge and self-efficacy following diagnosis and in the context of mild and moderate disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 40-80 years able to give written informed consent
* Confirmed diagnosis of mild or moderate COPD or diagnosed in the last 12 months with a confirmed diagnosis of COPD.
* FEV1 percent predicted value greater than 50% (Mild or Moderate COPD)
* Current or ex smoker
* FEV1/VC or FEV1/FVC Ratio less than 70%
* Currently taking inhaled medications
* Access to the internet at home, use of mobile technology and the ability to operate a web platform in English
* Consent to be contacted by phone, text and email.

Exclusion Criteria:

* FEV1 percent predicted less than 49% unless diagnosed in the last 12 months
* COPD exacerbation in the past 4 weeks
* Housebound patients
* Patients unable to read or use an internet enabled device.
* Alcohol and drug misuse
* Presence of a medical condition other than COPD which investigators feel would confound study outcome collection

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
COPD Assessment Test | 3 months
  This is a validated symptom scoring system used in COPD studies The CAT questionnaire contains eight questions and provides a reliable measure of the impact of COPD on health status. Patients read the two statements for each item, which describe the best and worst scenario, (e.g I never cough - I cough all the time), and decide where on the scale of 0-5 they fit. The maximum score is out of 40. The higher the CAT score the greater the impact of symptoms on their health status. Experts involved in the development of CAT suggest that any change of 2 or more in the patient's final score may indicate a clinically significant change. CAT will be recorded at the start prior to any intervention at visit one, at monthly telephone calls for the duration of the study and at end of study visit

SECONDARY OUTCOMES:
Incidence of treatment emergent Adverse and Serious Adverse Events (Safety and Tolerability) | 3 months
  Safety assessed by the incidence of treatment pathway emergent adverse event (AE's) and Serious Adverse Events (SAE's) at study completion. The number of adverse events and serious adverse events will be tabulated also by the number patients reporting an event.
Patient Activation Measurement (PAM) | 3 months
  PAM is a tool used for measuring the level of patient engagement in their healthcare. It was designed to assess an individual's knowledge, skill and confidence for self-management. PAM is a 13-item scale that asks people about their beliefs, knowledge and confidence for engaging in a wide range of health behaviours and then assigns an activation score based on their responses to the 13-item scale.
Health Economics Analysis | 3 months
  The measurement of health outcome used will be the Quality Adjusted Life Year (QALY) calculated using the EuroQol 5 Demension-5 Level questionnaire (EQ5D 5L).The EQ5D 5L is a validated questionnaire which comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Minimum score is 5 and maximum score is 25 patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' score maximum 100 and 'The worst health you can imagine score minimum 0.The use of NHS resources from an adjusted baseline period prior to staring the study compared to during the study will be used as a comparator for cost outcomes
Inhaler Technique | 3 months
  This will be assessed using the "7 Steps to successfully inhaler technique developed by the UK Inhaler Group. Each step is evaluated as being Good or Poor and the number of critical errors will be recorded.
Self Efficacy for Appropriate medication use Scale (SEAMS) | 3 months
  Seams is a validated medication adherence questionnaire. Designed to indicate level of self efficacy for medication management. The questionnaire contains 13 questions with 3 levels of response Not confident, Somewhat confident and very confident. The minimum score is 13 and maximum score 39. The higher the score indicates greater level of self efficacy
Change in Activity | 7 days post baseline and 7 days prior to end of study visit.
  Using FITBIT pedometers 12 patients from each arm will be allocated to activity monitoring to measure daily steps and improvement in total step count.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Wilkinson, Study Chair — my mhealth Ltd
Locations (1):
- my mhealth Limited, Bournemouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Callejas Gonzalez FJ, Genoves Crespo M, Cruz Ruiz J, Godoy Mayoral R, Agustin Martinez FJ, Martinez Garcia AJ, Tarraga Lopez PJ. UPLIFT study - understanding potential long-term impacts on function with tiotropium - and sub-analyses. Bibliographic resume of the obtained results. Expert Rev Respir Med. 2016 Sep;10(9):1023-33. doi: 10.1080/17476348.2016.1188693. Epub 2016 May 23. PMID 27176208
- [Background] Petty TL. The history of COPD. Int J Chron Obstruct Pulmon Dis. 2006;1(1):3-14. doi: 10.2147/copd.2006.1.1.3. PMID 18046898
- [Background] Lee SH, Kim KU, Lee H, Kim YS, Lee MK, Park HK. Factors associated with low-level physical activity in elderly patients with chronic obstructive pulmonary disease. Korean J Intern Med. 2018 Jan;33(1):130-137. doi: 10.3904/kjim.2016.090. Epub 2017 Jun 7. PMID 28602061
- [Result] WHO. (2008) COPD predicted to be third leading cause of death in 2030. [Online] Available at: http://www.who.int/respiratory/copd/World_Health_Statistics_2008/en/
- [Result] Crooks, MG. Thompson, J. Platten, S. Evans, C. Faruqi, S. (2017) P25 Living with COPD: a Public Awareness and Screening Campaign. BMJ Thorax. [Online] 72(3). Available at: http://thorax.bmj.com/content/72/Suppl_3/A94.3
- [Result] Lee HY, Choi SM, Lee J, Park YS, Lee CH, Kim DK, Lee SM, Yoon HI, Yim JJ, Kim YW, Han SK, Yoo CG. Effect of tiotropium on lung function decline in early-stage of chronic obstructive pulmonary disease patients: propensity score-matched analysis of real-world data. Int J Chron Obstruct Pulmon Dis. 2015 Oct 13;10:2185-92. doi: 10.2147/COPD.S91901. eCollection 2015. PMID 26508848
- [Result] Thabane M; COPD Working Group. Smoking cessation for patients with chronic obstructive pulmonary disease (COPD): an evidence-based analysis. Ont Health Technol Assess Ser. 2012;12(4):1-50. Epub 2012 Mar 1. PMID 23074432
- [Result] Arbillaga-Etxarri A, Gimeno-Santos E, Barberan-Garcia A, Benet M, Borrell E, Dadvand P, Foraster M, Marin A, Monteagudo M, Rodriguez-Roisin R, Vall-Casas P, Vilaro J, Garcia-Aymerich J; Urban Training Study Group. Socio-environmental correlates of physical activity in patients with chronic obstructive pulmonary disease (COPD). Thorax. 2017 Sep;72(9):796-802. doi: 10.1136/thoraxjnl-2016-209209. Epub 2017 Mar 1. PMID 28250201
- [Result] Waschki B, Kirsten A, Holz O, Muller KC, Meyer T, Watz H, Magnussen H. Physical activity is the strongest predictor of all-cause mortality in patients with COPD: a prospective cohort study. Chest. 2011 Aug;140(2):331-342. doi: 10.1378/chest.10-2521. Epub 2011 Jan 27. PMID 21273294
- [Result] Mantoani LC, Rubio N, McKinstry B, MacNee W, Rabinovich RA. Interventions to modify physical activity in patients with COPD: a systematic review. Eur Respir J. 2016 Jul;48(1):69-81. doi: 10.1183/13993003.01744-2015. Epub 2016 Apr 21. PMID 27103381